CLINICAL TRIAL: NCT01388010
Title: "Effect of the Consumption of a Fermented Dairy Product on Gastrointestinal Well-being in a Healthy Population of Women With Minor Digestive Symptoms"
Brief Title: Study of the Effect of a Fermented Dairy Product on Gastrointestinal Well Being in Adult Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NU325
Record Dates: First submitted 2011-07-03; First posted 2011-07-06 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Adult Women
Keywords: probiotics; gastrointestinal well being; digestive symptoms; healthy population

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 = Test product (Experimental): Arm 1 - Intervention 1 (probiotics)
  Interventions: Other: 1-Fermented Probiotic Dairy Product (test)
- 2 = Control product (Other): Arm 2 - Intervention 2 (control)
  Interventions: Other: 2-Milk-based non-fermented dairy product(control)

INTERVENTIONS:
Other: 1-Fermented Probiotic Dairy Product (test)
  Arms: 1 = Test product
Other: 2-Milk-based non-fermented dairy product(control)
  Arms: 2 = Control product

SUMMARY:
The purpose of this study is to evaluate the effect of a commercially available fermented dairy product containing probiotics (4 weeks, twice a day) on the improvement of gastrointestinal well being and digestive symptoms in adult women reporting minor digestive troubles among the general population.

ELIGIBILITY:
Inclusion Criteria:

* Female free-living subject aged from 18 to 60 years.
* Subject with a body mass index between 18 and 30.
* Subject with minor digestive symptoms as defined by screening questionnaire of frequency of digestive symptoms.
* Subject with normal stool frequency

Exclusion Criteria:

* Subject with a diagnosis of Irritable Bowel Syndrome (IBS) or other functional bowel disease (constipation, diarrhoea…)
* Subject with known organic disease, including an inflammatory bowel disease, a benign or malign tumour of intestine or colon and significant systemic disease
* Subject under prescription for medication for digestive symptoms such as anti-spasmodic, laxatives and anti-diarrheic drugs
* Subject having taken antibiotics in the last 4 weeks
* Pregnant subject or subject planning to become pregnant during the study; breast-feeding subject.
* Subject with known lactose intolerance or immunodeficiency
* Subject with known allergy to product component (milk protein for example)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 336 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- RPS Research France, Caen, France